CLINICAL TRIAL: NCT01308515
Title: A Comparative Clinical Evaluation of the Vanguard Knee System's Anterior Stabilized & Posterior Stabilized Tibial Bearings
Brief Title: Vanguard Knee Anterior Stabilized Versus Posterior Stabilized Bearing Study
Acronym: VGASPS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not find interested researchers/clinicians to complete study protocol.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 090809
Record Dates: First submitted 2010-06-02; First posted 2011-03-04 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis; Degenerative Arthritis
Keywords: knee; osteoarthritis; joint; replacement; knee surgery
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Posterior Stabilized (Other): Patients who received a PS (Posterior Stabilized) Tibial Bearing.
  Interventions: Device: Vanguard Knee System with PS Bearing
- Anterior Stablized (Other): Patients who received an AS (Anterior Stabilized) Tibial Bearing
  Interventions: Device: Vanguard Knee System with AS Bearing

INTERVENTIONS:
Device: Vanguard Knee System with AS Bearing — FDA cleared Tibial bearing that stabilizes the knee with an anterior lip, and is used with FDA cleared Vanguard CR (Cruciate Retaining) Femoral Component.
  Arms: Anterior Stablized
Device: Vanguard Knee System with PS Bearing — FDA cleared Tibial bearing that stabilizes the knee with a post that articulates with the FDA cleared Vanguard PS(Posterior Stabilizing) Femoral Component.
  Arms: Posterior Stabilized

SUMMARY:
The purpose of this study is to compare the performance of two FDA-cleared tibial bearings (replacement for cartilage in the knee) by collecting data on patients through 3 years of follow-up.

ELIGIBILITY:
Inclusion Criteria are identical to the indications stated in the FDA approved labeling for the device 510(k) K023546, K033489, and K050222. These indications are stated below:

* Painful and disabled knee joint resulting from osteoarthritis, rheumatoid arthritis, traumatic arthritis where one or more compartments are involved.
* Correction of varus, valgus, or posttraumatic deformity.
* Correction or revision of unsuccessful osteotomy, or arthrodesis.

Patient selection factors to be considered include:

* Need to obtain pain relief and improve function
* Ability and willingness of the patient to follow instructions, including control of weight and activity level
* A good nutritional state of the patient
* The patient must have reached full skeletal maturity

Exclusion criteria will be identical to the contraindications stated in the FDA approved labeling for the device 510(k) K023546, K033489, and K050222.

These contraindications are stated below:

-Absolute contraindications include: infection, sepsis, osteomyelitis, and failure of a previous joint replacement.

Relative contraindications include:

* Uncooperative patient or patient with neurologic disorders who are incapable of following directions
* Osteoporosis,
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Distant foci of infections which may spread to the implant site,
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram,
* Vascular insufficiency, muscular atrophy, neuromuscular disease,
* Incomplete or deficient soft tissue surrounding the knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Objective Knee Score | 1 Year Post-op
  Average objective knee score; includes a combination of range of motion and pain scores.

SECONDARY OUTCOMES:
Knee Society Score | 3 Years
  Average total knee score. Includes the objective and functional aspects of the knee score.
Dislocation | 3 Years
  Rate of Dislocation as reported by patients in a complication.
Survivorship | 3 Years
  Reports surivival of implant.
Reports of Radiographic Loosening via Complication Form | 3 Years
  A more specific survivorship element; will indicate rate of loosening if it occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Beres, MD, Study Director — Biomet (no investigators were selected for this study)